CLINICAL TRIAL: NCT04699110
Title: Efficacy of Intracoronary Adrenaline and Its Comparison With Intracoronary Adenosine in the Treatment of No-Reflow in Normotensive Patients With Acute Coronary Syndrome
Brief Title: Adrenaline for the Treatment of No-Reflow in Normotensive Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Cardiovascular Diseases, Pakistan (Other)
Responsible Party: Principal Investigator, Kamran Ahmed Khan, Assistant Professor of Cardiology, National Institute of Cardiovascular Diseases, Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERC-76/2020
Record Dates: First submitted 2021-01-05; First posted 2021-01-07 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Acute Coronary Syndrome; No-Reflow Phenomenon; Normotensive
MeSH Terms: conditions — Acute Coronary Syndrome; No-Reflow Phenomenon | interventions — Epinephrine; Adenosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental): Patients receiving intracoronary adrenaline
  Interventions: Drug: Adrenaline
- Control group (Active Comparator): Patients receiving intracoronary adenosine
  Interventions: Drug: Adenosine

INTERVENTIONS:
Drug: Adrenaline — Treatment group will receive adrenaline (100 to 400 mcg) for the treatment of No-reflow
  Arms: Treatment group
Drug: Adenosine — Control group will receive adenosine (100 to 400 mcg)
  Arms: Control group

SUMMARY:
No-reflow is defined as the lack of myocardial perfusion despite opening of the epicardial coronary vessels in the setting of percutaneous coronary intervention (PCI). It has been demonstrated that either impaired flow or the absence of flow is associated with an increased rate of mortality. Among available treatment options, intracoronary adenosine is widely used in clinical practice, moreover, adrenaline is a safe alternative for the cases where use of adenosine is limited due to presence of hypotension or bradycardia. Nonetheless, evidence from retrospective and observational studies suggest that intracoronary adrenaline is well tolerated and may exert encouraging effects in prompt recovery of flow in these patients. However, very limited data are available on efficacy of intracoronary (IC) adrenaline in normotensive patients. Therefore, this study is planned to study the hypothesis that; intracoronary adrenaline is safe and has significantly higher efficacy as compared to adenosine for the treatment of no-reflow in normotensive patients with acute coronary syndrome.

ELIGIBILITY:
Inclusion Criteria:

* All patients with acute coronary syndrome who developed No-reflow during PCI.
* Patients with systolic blood pressure of > 100 mmHg.

Exclusion Criteria:

* Hypotensive patients
* Patients with Valvular or congenital heart disease.
* Patients with Atypical chest pain
* Patients with Cardiomyopathy
* Patients with Pericarditis
* Patients with Myocarditis
* Patients refused to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Improvement in Thrombolysis in Myocardial Infarction (TIMI) flow grade | Immediately after administration of drug
Reduction in TIMI frame count | Immediately after administration of drug

SECONDARY OUTCOMES:
The major adverse cardiovascular events | During hospital stay and at 30-day follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Cardiovascular Diseases, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khan KA, Qamar N, Saghir T, Sial JA, Kumar D, Kumar R, Qayyum D, Yasin U, Jalbani J, Karim M. Comparison of Intracoronary Epinephrine and Adenosine for No-Reflow in Normotensive Patients With Acute Coronary Syndrome (COAR Trial). Circ Cardiovasc Interv. 2022 Feb;15(2):e011408. doi: 10.1161/CIRCINTERVENTIONS.121.011408. Epub 2022 Jan 10. PMID 35000456